CLINICAL TRIAL: NCT05996211
Title: The Swiss Neurodevelopmental Outcome Registry for Children With CHD
Acronym: SwissORCHID
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Lausanne Hospitals (Other); University of Geneva, Switzerland (Other); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Knirsch 02
Record Dates: First submitted 2023-07-18; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Neurodevelopmental Abnormality; Congenital Heart Disease; Cardiac Disease; Intensive Care Neurological Disorder
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Congenital heart disease (CHD) is the most frequent birth defect. As survival has significantly improved, attention has turned to neurodevelopmental outcomes of children undergoing heart surgery in early infancy. Since multiple risk factors contribute to neurodevelopmental alterations, a nationwide registry collecting data on medical characteristics, interventions, clinical course and neurodevelopment until school-age is needed to improve the quality of management, identify risk- and protective factors affecting neurodevelopment, and facilitate multicenter trials.

Methods and analysis: The Swiss Outcome Registry for CHIldren with severe congenital heart Disease (ORCHID) is a nationwide, prospective, population-based patient registry developed (1) to collect baseline characteristics and clinical data of CHD patients operated with bypass-surgery or hybrid procedures in the first 6 weeks of life in Switzerland, (2) to monitor long-term neurodevelopment, and (3) to relate clinical characteristics and neurodevelopment to identify risk and protective factors in these children. This registry started data collection relating to pregnancy, birth, preoperative course, catheter-based and surgical treatment, postoperative course and reinterventions in 2019. The primary outcome includes standardised neurodevelopmental assessments at 9 to 12 months, 18 to 24 months and 5.5 to 6 years. Investigators expect to include 80 to 100 children per year. Correlation and regression analyses will be used to investigate risk- and protective factors influencing neurodevelopment.

Ethics and dissemination of results: Swiss ORCHID received support by the Accentus Charitable Foundation, the Anna Mueller Grocholoski Foundation, the Swiss Society of Pediatric Cardiology, and the Corelina - Foundation and was approved by the cantonal ethics committees. Findings will be presented at national and international scientific meetings, and published in peer-reviewed journals. Results will also be shared with patient organizations, primary health care providers, and public health stakeholders to ensure a widespread dissemination of the results.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (including preterm born children) with severe CHD
* Requiring an invasive cardiac intervention (including heart-lung-machine) within the first 6 weeks of life.

Exclusion Criteria:

* Neonates (including preterm born children) with simple CHD
* Requiring simple cardiac surgery or catheter intervention such as closure of patent arterial duct or simple repair of aortic coarctation without heart-lung-machine and low impact on neurodevelopmental outcome.

Ages: 1 Week to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with severe CHD
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Bayley scales of infant and toddler development III at one year of age | One year of age
  Neurodevelopmental outcome measurement at one year of age (normal value 100, higher values mean better outcome)
Bayley scales of infant and toddler development III at two years of age | Two years of age
  Neurodevelopmental outcome measurement at two years of age (normal value 100, higher values mean better outcome)
Bayley scales of infant and toddler development III at five years of age | Five years of age
  Neurodevelopmental outcome measurement at five years of age (normal value 100, higher values mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Knirsch, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (3):
- Switzerland (3):
  - University of Bern, Bern
  - University of Lausanne, Lausanne
  - University Children's Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Natterer J, Schneider J, Sekarski N, Rathke V, Adams M, Latal B, Borradori-Tolsa BT, Bouhabib M, Fuhrer Kradolfer K, Glockler M, Hutter D, Kelly J, L'Ebraly C, Pfluger MR, Polito A, von Rhein M, Knirsch W. ORCHID (Outcome Registry for CHIldren with severe congenital heart Disease) a Swiss, nationwide, prospective, population-based, neurodevelopmental paediatric patient registry: framework, regulations and implementation. Swiss Med Wkly. 2022 Sep 2;152:w30217. doi: 10.4414/smw.2022.w30217. eCollection 2022 Aug 29. PMID 36074038
- [Derived] Knirsch W, De Silvestro A, Rathke V, L'Ebraly C, Natterer JC, Schneider J, Sekarski N, Latal B, Borradori-Tolsa C, Bouhabib MS, Fuhrer Kradolfer K, Glockler M, Hutter D, Pfluger MR, Kaiser L, Polito A, Kelly-Geyer JF, von Rhein M; Swiss ORCHID group. Impact of postoperative necrotizing enterocolitis after neonatal cardiac surgery on neurodevelopmental outcome at 1 year of age. Front Pediatr. 2024 Aug 6;12:1380582. doi: 10.3389/fped.2024.1380582. eCollection 2024. PMID 39165487
- See also: Publication of Swiss ORCHID — https://pubmed.ncbi.nlm.nih.gov/?term=%22Swiss+medical+weekly%22%5BJournal%5D+AND+2022%2F9%2F2%5BDate+-+Publication%5D